CLINICAL TRIAL: NCT05568433
Title: New Biomarkers in the Intracystic Liquid of Cystic Pancreatic Lesions
Brief Title: New Biomarkers in the Intracystic Liquid of Inflammatory and Non-inflammatory Pancreatic Cysts
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Olar Miruna-Patricia, Principal Investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: 202042018
Record Dates: First submitted 2022-09-25; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cyst
Keywords: pancreatic cyst; EUS-FNA; intracystic fluid
MeSH Terms: conditions — Pancreatic Cyst | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, cystic fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound fine needle aspiration (EUS-FNA) — Patients with pancreatic cysts who underwent endoscopic ultrasound and endoscopic fine needle aspiration for diagnostic and therapeutic purpose. A sample of the cyst fluid and frozen serum was collected from the patients and stored at minus 80 degrees.
  Other Names: ELISA measurements of cystic fluid

SUMMARY:
Due to the advances made in the field of the imaging techniques and their common use, pancreatic cysts are more and more incidentally found.

Pancreatic pseudocysts can be misdiagnosed as cystic neoplasms, in particular when there is no clinical history of acute or chronic pancreatitis. Pancreatic cystic neoplasms on the other hand are rare, but are difficult to diagnose accurately.

Neutrophil gelatinase-associated lipocalin (NGAL) , interleukin 1 Beta (IL1beta) and High Mobility Group AT-Hook 2 (HmgA2) are molecules implicated in the process of inflammation and tumour development. The diagnostic value of their concentration in pancreatic cysts is not established yet.

Study aim to asses the significance of NGAL,IL1Beta and HMGA2 concentration in cystic fluid obtained by endoscopic ultrasound (EUS) with EUS-guided fine-needle aspiration (EUS-FNA) and serum level for discriminating between inflammatory and non-inflammatory pancreatic cyst.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-90 years with an unclear specific diagnosis of pancreatic cysts
* pancreatic cyst >15mm on CT or MRI
* patients with pseudocysts with indication for drainage

Exclusion Criteria:

* refusal to participate
* platelet level < 50000/mm3 and International normalized ratio (INR >1.5)
* duodenal stenosis
* severe chronic pancreatitis
* history of pancreatic cancer or major upper abdominal surgery
* congestive heart failure
* the liquid sample < 1ml;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged 18-90 years diagnosed with an unclear specific diagnosis of pancreatic cysts >15mm on Computer tomography scan (CT) or Magnetic resonance imaging (MRI) and patients with pseudocysts with indication for drainage , admitted to our hospital (the Regional Institute of Gastroenterology and Hepatology in Cluj-Napoca, Romania)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Role of the cyst fluid concentrations of the specific biomarkers for differentiation the pancreatic cystic lesions | through study completion, an average of 1 year
  Measurement the cyst fluid concentration of NGAL, IL1beta, HMGA2, expressed in nanograms/dl

SECONDARY OUTCOMES:
The Correlation between cyst fluid concentration and serum level of the specific biomarkers | through study completion, an average of 1 year
  coefficient of correlation between the two values

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Seicean, Professor, Study Director — Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Locations (1):
- Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan JH, Chin W, Shaikh AL, Zheng S. Pancreatic pseudocyst: Dilemma of its recent management (Review). Exp Ther Med. 2021 Feb;21(2):159. doi: 10.3892/etm.2020.9590. Epub 2020 Dec 18. PMID 33456526
- [Background] Del Chiaro M, Segersvard R, Pozzi Mucelli R, Rangelova E, Kartalis N, Ansorge C, Arnelo U, Blomberg J, Lohr M, Verbeke C. Comparison of preoperative conference-based diagnosis with histology of cystic tumors of the pancreas. Ann Surg Oncol. 2014 May;21(5):1539-44. doi: 10.1245/s10434-013-3465-9. Epub 2014 Jan 3. PMID 24385209
- [Background] van Huijgevoort NCM, Del Chiaro M, Wolfgang CL, van Hooft JE, Besselink MG. Diagnosis and management of pancreatic cystic neoplasms: current evidence and guidelines. Nat Rev Gastroenterol Hepatol. 2019 Nov;16(11):676-689. doi: 10.1038/s41575-019-0195-x. Epub 2019 Sep 16. PMID 31527862
- [Background] Chakraborty S, Kaur S, Guha S, Batra SK. The multifaceted roles of neutrophil gelatinase associated lipocalin (NGAL) in inflammation and cancer. Biochim Biophys Acta. 2012 Aug;1826(1):129-69. doi: 10.1016/j.bbcan.2012.03.008. Epub 2012 Mar 31. PMID 22513004
- [Background] Clerico A, Galli C, Fortunato A, Ronco C. Neutrophil gelatinase-associated lipocalin (NGAL) as biomarker of acute kidney injury: a review of the laboratory characteristics and clinical evidences. Clin Chem Lab Med. 2012 Feb 15;50(9):1505-17. doi: 10.1515/cclm-2011-0814. PMID 22962216
- [Background] Devarajan P. Neutrophil gelatinase-associated lipocalin--an emerging troponin for kidney injury. Nephrol Dial Transplant. 2008 Dec;23(12):3737-43. doi: 10.1093/ndt/gfn531. Epub 2008 Sep 22. No abstract available. PMID 18809975
- [Background] Bhatia R, Muniyan S, Thompson CM, Kaur S, Jain M, Singh RK, Dhaliwal A, Cox JL, Akira S, Singh S, Batra SK, Kumar S. Neutrophil Gelatinase-Associated Lipocalin Protects Acinar Cells From Cerulein-Induced Damage During Acute Pancreatitis. Pancreas. 2020 Nov/Dec;49(10):1297-1306. doi: 10.1097/MPA.0000000000001690. PMID 33122517
- [Background] Chakraborty S, Kaur S, Muddana V, Sharma N, Wittel UA, Papachristou GI, Whitcomb D, Brand RE, Batra SK. Elevated serum neutrophil gelatinase-associated lipocalin is an early predictor of severity and outcome in acute pancreatitis. Am J Gastroenterol. 2010 Sep;105(9):2050-9. doi: 10.1038/ajg.2010.23. Epub 2010 Feb 23. PMID 20179686
- [Background] Santiago-Sanchez GS, Pita-Grisanti V, Quinones-Diaz B, Gumpper K, Cruz-Monserrate Z, Vivas-Mejia PE. Biological Functions and Therapeutic Potential of Lipocalin 2 in Cancer. Int J Mol Sci. 2020 Jun 19;21(12):4365. doi: 10.3390/ijms21124365. PMID 32575507
- [Background] Kaur S, Baine MJ, Guha S, Ochi N, Chakraborty S, Mallya K, Thomas C, Crook J, Wallace MB, Woodward TA, Jain M, Singh S, Sasson AR, Skinner V, Raimondo M, Batra SK. Neutrophil gelatinase-associated lipocalin, macrophage inhibitory cytokine 1, and carbohydrate antigen 19-9 in pancreatic juice: pathobiologic implications in diagnosing benign and malignant disease of the pancreas. Pancreas. 2013 Apr;42(3):494-501. doi: 10.1097/MPA.0b013e31826a8597. PMID 23146921